CLINICAL TRIAL: NCT05621005
Title: Rifaximin Prophylaxis Against Recurrence of Spontaneous Bacterial Peritonitis and Occurrence of Hepatorenal Syndrome in Decompensated Cirrhotic Egyptian Patients
Brief Title: Rifaximin Prophylaxis for Spontaneous Bacterial Peritonitis and Hepatorenal Syndrome in Cirrhotic Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Samar Atef Sebaweh Mohammed (Other)
Responsible Party: Sponsor-Investigator, Samar Atef Sebaweh Mohammed, assistant lecturer, Ain Shams University
Organization: Ain Shams University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: SBP prophylaxis
Record Dates: First submitted 2022-11-12; First posted 2022-11-17 (Actual); Last update posted 2022-11-21 (Actual); Status verified 2022-11

CONDITIONS: Ascites Infection
Keywords: Rifaximin; Norflixacin; Spontaneous bacterial peritonitis
MeSH Terms: interventions — Rifaximin

STUDY DESIGN:
Intervention Model Description: Study design: non inferiority prospective non randomized controlled trial
  Study population and setting:
  The study enrolled patients with chronic liver disease and ascites who were monitored at outpatient clinics or who were admitted to Ain Shams University hospitals.
  Sample size: 104 patients with decompensated liver cirrhosis were enrolled in the study. The Control Group (n=52), to receive standard of care treatment & Norfloxacin prophylaxis for the decompensated liver disease and a second Treatment Group (n=52) who will receive Rifaximin prophylaxis in addition to the original management.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- treatment group or Rifaximin group (Experimental): they received Rifaximin 550 milligram every 12 hour
  Interventions: Drug: Rifaximin 550 milligram Oral Tablet [XIFAXAN]
- control group or Norfloxacin group (Active Comparator): they received Norfloxacin 400 milligram per day
  Interventions: Drug: Rifaximin 550 milligram Oral Tablet [XIFAXAN]

INTERVENTIONS:
Drug: Rifaximin 550 milligram Oral Tablet [XIFAXAN] — Rifaximin was given on dose of 550 milligram every 12 hours orally for at least 3 months
  Other Names: xifaxan

SUMMARY:
Norfloxacin is the most commonly used drug for the prophylaxis against spontaneous bacterial peritonitis (SBP) in patients with liver cirrhosis. Rifaximin, another broad spectrum antibiotic with only trivial absorption from the gut, is used for the treatment of traveler's diarrhea and prevention of hepatic encephalopathy.

DETAILED DESCRIPTION:
Prophylaxis against spontaneous bacterial peritonitis (SBP) in cirrhotic patients recovered from an episode of SBP using Norfloxacin 400 mg/day is currently established standard of care. Recently we are facing the growing challenge of standard SBP prophylaxis lacking efficacy as extended spectrum beta-lactamases and fluoro-quinolone resistant bacteria in isolates of patients on Norfloxacin.

Prophylaxis against Hepatorenal Syndrome in decompensated liver cirrhosis is limited to IV administration of Albumin in patients who develop SBP and the prevention of SBP using Norfloxacin.

this study aims to investigate the effectiveness of Rifaximin in decompensated cirrhotic patients against SBP as a secondary prophylaxis measure and Hepatorenal Syndrome.

our study was non inferiority prospective non randomized controlled trial The study enrolled patients with chronic liver disease and ascites who were monitored at outpatient clinics or who were admitted to Ain Shams University hospitals.104 patients with decompensated liver cirrhosis were enrolled in the study, The Control Group (n=52), to receive standard of care treatment & Norfloxacin prophylaxis for the decompensated liver disease and a second Treatment Group (n=52) who will receive Rifaximin prophylaxis in addition to the original management.

ELIGIBILITY:
Inclusion Criteria:

1. Decompensated cirrhotic patients (Child B or C, ascetic patients).
2. Adult male/female aged >18 years old.
3. History or evidence of previous attack of SBP and currently clinically free from SBP.

Exclusion Criteria:

1. Recent abdominal surgery.
2. Patients with renal impairment (serum creatinine >1.5mg/dl) at baseline.
3. Patients on renal replacement therapy (RRT) at baseline.
4. Sonographic evidence of Nephropathy other than grade I nephropathy in ascetic patients
5. intraabdominal source of infection (e.g. intra-abdominal abscesses, cholecystitis or acute pancreatitis).
6. Patients with current evidence of upper Urinary tract infection.
7. Other comorbidities affecting the patient survival e.g. significant cardiac disease, pulmonary disease, portal vein thrombosis, hepatocellular carcinoma or other malignancies, etc.
8. Sepsis.
9. Current or recent treatment with nephrotoxic drugs or contrast material injection.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2022-08-01 (Actual)

PRIMARY OUTCOMES:
secondary prophylaxis of SBP and primary prophylaxis for hepatorenal syndrome | 3 months
  our study was conducted to test the efficacy of Rifaximin in prevention of recurrence of SBP and occurrence of hepatorenal syndrome

CONTACTS AND LOCATIONS:
Overall Officials: Samar A Sebaweh, master, Principal Investigator — assistant lecturer
Locations (1):
- faculty of medicine Ain Shams university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
individual participant data will be shared including inclusion criteria and the final statical results
Supporting Information: Study Protocol
Time Frame: 3 to 5 months
Access Criteria: through the official e mail and the publishing journal

REFERENCES:
- [Background] Acevedo JG, Cramp ME. Hepatorenal syndrome: Update on diagnosis and therapy. World J Hepatol. 2017 Feb 28;9(6):293-299. doi: 10.4254/wjh.v9.i6.293. PMID 28293378
- [Background] Dong T, Aronsohn A, Gautham Reddy K, Te HS. Rifaximin Decreases the Incidence and Severity of Acute Kidney Injury and Hepatorenal Syndrome in Cirrhosis. Dig Dis Sci. 2016 Dec;61(12):3621-3626. doi: 10.1007/s10620-016-4313-0. Epub 2016 Sep 21. PMID 27655104
- [Background] Fernandez J, Tandon P, Mensa J, Garcia-Tsao G. Antibiotic prophylaxis in cirrhosis: Good and bad. Hepatology. 2016 Jun;63(6):2019-31. doi: 10.1002/hep.28330. Epub 2016 Jan 11. PMID 26528864
- [Background] Moreau R, Elkrief L, Bureau C, Perarnau JM, Thevenot T, Saliba F, Louvet A, Nahon P, Lannes A, Anty R, Hillaire S, Pasquet B, Ozenne V, Rudler M, Ollivier-Hourmand I, Robic MA, d'Alteroche L, Di Martino V, Ripault MP, Pauwels A, Grange JD, Carbonell N, Bronowicki JP, Payance A, Rautou PE, Valla D, Gault N, Lebrec D; NORFLOCIR Trial Investigators. Effects of Long-term Norfloxacin Therapy in Patients With Advanced Cirrhosis. Gastroenterology. 2018 Dec;155(6):1816-1827.e9. doi: 10.1053/j.gastro.2018.08.026. Epub 2018 Aug 23. PMID 30144431
- [Background] Soriano G, Guarner C, Teixido M, Such J, Barrios J, Enriquez J, Vilardell F. Selective intestinal decontamination prevents spontaneous bacterial peritonitis. Gastroenterology. 1991 Feb;100(2):477-81. doi: 10.1016/0016-5085(91)90219-b. PMID 1985045
- [Background] Vlachogiannakos J, Viazis N, Vasianopoulou P, Vafiadis I, Karamanolis DG, Ladas SD. Long-term administration of rifaximin improves the prognosis of patients with decompensated alcoholic cirrhosis. J Gastroenterol Hepatol. 2013 Mar;28(3):450-5. doi: 10.1111/jgh.12070. PMID 23216382